CLINICAL TRIAL: NCT06815510
Title: Multicentral Observational Prospective Study on Prevalence of Post Anesthesia Care Unit Complications and Associated Factors
Brief Title: Prevalence of Post Anesthesia Care Unit Complications and Associated Factors
Status: Recruiting | Type: Observational
Sponsor: Ángel Becerra-Bolaños, MD PhD (Other)
Collaborators: Mekelle University (Other); Jimma University (Other); Haramaya Unversity (Other)
Responsible Party: Sponsor-Investigator, Ángel Becerra-Bolaños, MD PhD, Principal Investigator, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Other Study IDs: MU-IRB 2418/2024
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Care; Complications of Surgical Procedures or Medical Care; Inpatients; Ethiopia; Multicenter Prospective Study
Keywords: postoperative complications; postanesthesia care unit
MeSH Terms: conditions — Postoperative Complications | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients admitted to the postanesthesia care unit: Adult patients admitted to the postanesthesia care unit following surgery under general, regional, or monitored anesthesia
  Interventions: Diagnostic Test: Questionnaire and Physical Exam

INTERVENTIONS:
Diagnostic Test: Questionnaire and Physical Exam — Patients will be followed up to find out any of these complications: pulmonary, hemodynamic complications, temperature disturbances, or pain
  Other Names: Postoperative complications in the PACU

SUMMARY:
The post-anesthesia care unit (PACU) is a crucial component of the surgical process, providing patients with vital support and monitoring as they recover from anesthesia. Despite advancements in perioperative anesthesia, PACU complications are still common. PACU organization and setup in low-income country like Ethiopia is poor. Previous research's done in some neighbor African countries presumed to have comparable to sociodemographic and economical profile shows varied degree of incidence and prevalence of PACU complication and associated factors. The main objective of this study is to determine the prevalence of PACU complications and its associated factors.

An institutional based prospective cohort study will be conducted in the PACUs of the three selected tertiary care hospitals in Ethiopia from Februery 15, 2025 to June 30, 2025. These data will be compared with those obtained in a tertiary hospital in Spain.

DETAILED DESCRIPTION:
Studying the prevalence and associated factors of PACU complications will be of great academic importance, serving as a valuable reference and resource for further research. It will also help identify risk factors attributable to PACU complications, providing critical insights for hospital administrators and policymakers in making informed decisions about resource allocation and system design to minimize these complications. Understanding the prevalence and potential risk factors of PACU complications is essential for optimizing patient care and improving outcomes. Identified risk factors for postoperative complications in the PACU include female sex, longer duration of anesthesia, and the occurrence of intraoperative complications. This study aims to explore the prevalence of complications in the PACU and identify potential contributing factors, providing valuable insights for healthcare providers and policymakers seeking to improve PACU care. the potential significance and implications of the study findings, includes; Improving the understanding of PACU complications and the associated risk factors, informing the development of targeted prevention and management strategies, enhancing patient safety and quality of care in the perioperative setting and providing a basis for future research and evidence-based clinical guidelines. The study will involve surgical patients admitted to the Post-Anesthesia Care Units (PACUs) of four hospitals: Hiwot Fana Comprehensive Specialized Hospital, Ayder Comprehensive Specialized Hospital, Jimma University Medical Center (Ethiopia) and Hospital Universitario de Gran Canaria Doctor Negrín (Spain). The research will take place from February 15, 2025, to June 30, 2025. Multicenter, prospective, observational cohort study will be conducted reviewing patients admitted to the PACU. Analyzing complications in all patients admitted to the PACUs at the four selected hospitals following surgery under general, regional, or monitored anesthesia will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the Post-Anesthesia Care Units (PACUs) following surgery under general, regional, or monitored anesthesia

Exclusion Criteria:

* Patients who are taken directly to the ICU, ward, discharged, or transferred immediately after surgery.
* Patients who do not provide informed consent for enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the Post-Anesthesia Care Units (PACUs) following surgery under general, regional, or monitored anesthesia who have signed the informed consent preoperatively will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1532 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with postoperative complications in the postanesthesia care unit | 8 postoperative hours
  Patients will be followed up during their stay in the PACU looking for the appearance of respiratory and hemodynamic complications, temperature disturbances or pain

CONTACTS AND LOCATIONS:
Overall Officials: Ataklti Adhanom, MD, Principal Investigator — Mekelle University; Sirak Worku, MD, Principal Investigator — Haramaya University; Badhaasaa Beyene, MD, Principal Investigator — Haramaya University; Ruth Desta, MD, Principal Investigator — Haramaya University; Edosa Kejela, MD, Principal Investigator — Jimma University; Ángel Becerra-Bolaños, MD PhD, Principal Investigator — Hospital Universitario de Gran Canaria Doctor Negrín; Fekrey Berhe Gebru, MD, Principal Investigator — Mekelle University; Frtuna Zeray, MD, Principal Investigator — Mekelle University; Aemero Awoke, MD, Principal Investigator — Jimma University; Teklay Tesfay, MD, Principal Investigator — Mekelle University
Locations (4):
- Ethiopia (3):
  - Haramaya University, Harar
  - Jimma University, Jimma
  - Mekelle University, Mek'ele
- Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria, Spain

IPD SHARING:
Plan to Share IPD: Undecided
IPD used in the results publication will be shared.